CLINICAL TRIAL: NCT02665676
Title: Embryonal Tumors of Infancy & Childhood: South Egypt Cancer Institute Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Ped Embryonal Tumors SECI
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms, Embryonal; Embryonal Neoplasms
Keywords: Childhood Cancer; Pediatric Oncology; Embryonal Neoplasms; Embryonic Neoplasms; Embryonic Tumors; Embryonal Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate demographic & disease characteristics of pediatric cancer patients diagnosed with one of embryonal tumors to identify the prevalence, the spectrum of these disease entities & treatment outcomes in these patients.

DETAILED DESCRIPTION:
Background:

Embryonal tumors arise from cells that are normally present in the developing embryo and originate in developing tissues and organ systems. These tumors occur almost exclusively in children, and are usually diagnosed in children before age 5 years.

The group is heterogeneous and includes relatively common pediatric tumors as well as rare tumors. Three common types of embryonal tumors in children are neuroblastoma, Wilms tumor (WT), and retinoblastoma. Other embryonal tumors, include medulloblastoma and rhabdomyosarcoma.

Patients & Methods:

From January 2001 to December 2015, retrieval & analysis of the medical records of pediatric patients with embryonal tumors will be made at the pediatric oncology department, South Egypt Cancer Institute which represents the largest referral center in Upper Egypt. These data will be categorized according to demographic characteristics, clinico-pathologic features, treatment modalities received, and outcomes of treatments in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than or equal to 18 years.
* Patients diagnosed with any of embryonal neoplasms.

Exclusion Criteria:

• Patients whose age more than 18 years.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with any of embryonal neoplasms, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Tulla M, Berthold F, Graf N, Rutkowski S, von Schweinitz D, Spix C, Kaatsch P. Incidence, Trends, and Survival of Children With Embryonal Tumors. Pediatrics. 2015 Sep;136(3):e623-32. doi: 10.1542/peds.2015-0224. PMID 26304823
- [Background] Ward E, DeSantis C, Robbins A, Kohler B, Jemal A. Childhood and adolescent cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):83-103. doi: 10.3322/caac.21219. Epub 2014 Jan 31. PMID 24488779